CLINICAL TRIAL: NCT01418495
Title: Pharmacokinetics of the Chimeric Anti-GD2 Antibody, ch14.18, in Children With High-Risk Neuroblastoma
Brief Title: Pharmacokinetics of Ch14.18 in Younger Patients With High-Risk Neuroblastoma
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCI-2011-02975; NCI-2011-02975 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CHP-1002; CDR0000701215; CHP1002 (Other: Children's Hospital of Philadelphia); 9122 (Other: CTEP); P30CA016520 (NIH)
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Localized Resectable Neuroblastoma; Localized Unresectable Neuroblastoma; Neurotoxicity Syndrome; Pain; Regional Neuroblastoma; Stage 4 Neuroblastoma; Stage 4S Neuroblastoma
MeSH Terms: conditions — Neurotoxicity Syndromes; Pain; Neuroblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood

GROUPS / COHORTS (1):
- Ancillary-Correlative (pharmacokinetics of ch14.18): Patients undergo blood sample collection at baseline and during and after course 1, 3, or 5 of treatment for pharmacokinetic analysis. Some patients undergo blood sample collection at baseline and during and after two treatment courses (1 and 3, 1 and 5, or 3 and 5).
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Pharmacological Study

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Correlative studies
  Other Names: Cytologic Sampling
Other: Pharmacological Study — Correlative studies

SUMMARY:
This research trial is studying how Ch14.18 acts in the body of younger patients with high-risk neuroblastoma. Studying samples of blood from patients with cancer receiving Ch14.18 may help doctors learn more about how this drug is used by the body to develop better ways to give the drug to potentially improve its effectiveness and lessen its side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Describe the pharmacokinetics of ch14.18 (monoclonal antibody Ch14.18) in children with high-risk neuroblastoma.

II. Quantify the degree of inter-patient and intra-patient variability in the clearance of ch14.18, and correlate ch14.18 clearance with patient characteristics, the presence of human anti-chimeric antibody (HACA), tumor burden (assessed on scans), and plasma GD2 levels to identify sources of variability in the clearance.

III. Develop a pharmacokinetic model to describe the pharmacokinetic profile of ch14.18 and derive pharmacokinetic (PK) parameters.

SECONDARY OBJECTIVES:

I. Correlate plasma concentrations of ch14.18 with the severity of neuropathic pain, which is being quantified using an observational pain scale, and the total dose of morphine administered to control pain.

II. Develop a limited sampling strategy that will accurately quantify the area under the curve (AUC) of ch14.18.

III. Simulate alternative dosing strategies with the pharmacokinetic model in order to reduce variability and simplify drug administration.

OUTLINE:

Patients undergo blood sample collection at baseline and during and after course 1, 3, or 5 of treatment for pharmacokinetic analysis. Some patients undergo blood sample collection at baseline and during and after two treatment courses (1 and 3, 1 and 5, or 3 and 5).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of high-risk neuroblastoma
* Enrolled on the COG protocol ANBL0032 or ANBL0931 and eligible to receive ch14.18 according to the criteria on these primary treatment protocols
* Parental informed consent and verbal assent of the subject when appropriate

Exclusion Criteria:

* Prior testing demonstrating the presence of HACA
* Anaphylactic reaction to ch14.18 on a prior treatment cycle

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with high-risk neuroblastoma enrolled on Children's Oncology Group (COG) ANBL0032 or ANBL0931
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2011-05-26 (Actual)

PRIMARY OUTCOMES:
PK parameters of monoclonal antibody ch14.18 in children with high?risk neuroblastoma during and after 4 daily 10?hour infusions | Before and after infusion on days 3-5; before, after, 4-6 hours after, and 12-14 hours after infusion on day 6; on the morning of days 10, 14, 17, and 24; and before infusion on day 31
  PK parameters include the peak concentration, trough concentration, AUC, clearance, volume of distribution, half-life, and mean residence time. PK parameters will be derived from the plasma concentration-time data. A one-compartment model fit to the concentration-time data will estimated the volume of distribution and the first order elimination rate constant, which will in turn be used to calculate clearance, half-life, AUC0-infinity, AUC0-last, and the mean residence time. An error function and the dependency for each fitted parameter will be reported.
Coefficient of variation of monoclonal antibody ch14.18 clearance | Up to 58 days
  The coefficient of variation of Ch14.18 clearance is used to quantify the degree of inter-patient and intra-patient variability of monoclonal antibody ch14.18 pharmacokinetics. The relationship between patient characteristics, HACA, tumor burden, and plasma GD2 levels will be assessed graphically in an exploratory fashion with regression models.

SECONDARY OUTCOMES:
Severity of neuropathic pain, quantified using an observational pain scale based on the Face, Legs, Activity, Cry, Consolability scale (FLACC) and the total dose of morphine delivered | Up to 58 days
  The pain measures will be correlated with plasma concentrations of monoclonal antibody ch14.18 simulated using the PK model and the monoclonal antibody ch14.18 AUC0-96 hours. The overall drug exposure during the infusion will be correlated with the total morphine dose administered over the 4 days of treatment.
AUC of Ch14.18 | Up to 58 days
  A limited sampling strategy that will accurately quantify the AUC of monoclonal antibody ch14.18 will be developed.
Alternative dosing strategies | Up to 58 days
  Alternative dosing strategies will be simulated with the pharmacokinetic model in order to reduce variability and simplify drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Frank M Balis, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States